CLINICAL TRIAL: NCT04909918
Title: The Impact of Dexamethasone Versus Methylprednisolone Upon Neutrophil/Lymphocyte Ratio (NLR) in COVID-19 Diseased Patients Admitted in ICU
Brief Title: Impact of Steroids on Inflammatory Response in Covid-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300610
Record Dates: First submitted 2021-05-30; First posted 2021-06-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone; Calcium Dobesilate; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group D )Dexamethasone (Experimental): Intravenous dexamethasone 8 mg/day given for 7 days
  Interventions: Drug: Dexamethasone
- (Group M) methylprednisolone (Experimental): Intravenous methylprednisolone 1 mg/kg/day in 2 divided doses per day given for 7 days
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone — Baseline laboratory & clinical data will be taken before and after the study drugs according to our protocol.Intravenous dexamethasone 8 mg/day given for 7 days
  Other Names: Decadron
  Arms: (Group D )Dexamethasone
Drug: Methylprednisolone — Baseline laboratory & clinical data will be taken before and after the study drugs according to our protocol. Intravenous methylprednisolone 1 mg/kg/day in 2 divided doses per day given for 7 days
  Other Names: Solu-medrol
  Arms: (Group M) methylprednisolone

SUMMARY:
we designed this study to observe the efficacy and safety of dexamethasone versus methylprednisolone in covid-19 diseased patients upon monitoring the inflammatory response and to compare the outcome when these steroids will be given in covid-19 diseased patients in our ICU.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients or their relatives. The study will involve adults (age 18-no limit years) who will be diagnosed covid-19 with destructive inflammatory immune response needing ICU admission to be run on steroid therapy.

Patients will be assigned randomly to two groups (30 subjects each). The study drug will be delivered in opaque bags labeled "study drug" and in (Group D) intravenous dexamethasone 8 mg/day given for 7 days, in (Group M) intravenous methylprednisolone 1 mg/kg/day in 2 divided doses per day given for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-no limit years) who will be diagnosed covid-19
* With destructive inflammatory immune response needing ICU admission to be run on steroid therapy.

Exclusion Criteria:

* Severe immunosuppression like HIV (Human immunodeficiency Virus)
* Long term use of immunosuppressant for any other chronic illness
* Pregnant or lactating females
* Patients who are on chronic use of corticosteroids like asthma, rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Neutrophil/lymphocyte ratio (NLR) | 7 days
  Monitoring of systemic inflammation by follow up of neutrophil/lymphocyte ratio (NLR) at days 0, 48 hour, 72 hour and at day 7 between the two study drugs

SECONDARY OUTCOMES:
Interleukin-6 (IL-6) level | 7days
  Serum level of IL-6 is taken before start drug study &at 7 days to assess inflammatory and immune response
C-reactive protein (CRP) test | 3 days
  CRP test is done before start drug study, at 48hour and 72 hour to assess inflammatory response
Arterial oxygen tension/ inspired oxygen fraction (P/F ratio) | 3 days
  Assessing p/f ratio from arterial blood gas to monitor oxygenation & need for upgrading of oxygen, this is monitored before start of study drugs,at 48 hour and 72 hour
ICU stay | 7 days
  Period of patients admission in the ICU
ICU mortality | 7days
  Short-term icu mortality (7 days) for patients will be expired

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polidoro RB, Hagan RS, de Santis Santiago R, Schmidt NW. Overview: Systemic Inflammatory Response Derived From Lung Injury Caused by SARS-CoV-2 Infection Explains Severe Outcomes in COVID-19. Front Immunol. 2020 Jun 26;11:1626. doi: 10.3389/fimmu.2020.01626. eCollection 2020. PMID 32714336